CLINICAL TRIAL: NCT03091283
Title: A Survey Study of Time Management in Nurse Anaesthetist Students
Brief Title: Time Management in Nurse Anaesthetist Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Suchittra Bumrongsawat, Miss, Siriraj Hospital
Other Study IDs: Si 088/2017
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Educational Problems
Keywords: time management, anaesthesia training program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nurse anaesthetist student is a registered nurse who spends 1- year training in anaesthesia, has to work laboriously to cope with all assigned activities day and night. Time management, therefore, becomes a practical tool for nurse student to reach her goal. However, many factors act as barriers to nurse students' attaining and maintaining a high grade point average (GPA). Investigators would like to determine the effect of skills in time management on GPA amongst faculty nursing students.

DETAILED DESCRIPTION:
Skills in time management are crucial for academic success. It can be defined as clusters of behavioural set that are essentials in the organisation of learning load. These are comprised of activities such as planning, prioritising, preparation, and following schedules. Consequently, it yields an impact on students' achievement.

Nurse anaesthetist student is a registered nurse who spends 1- year training in anaesthesia. She has to work laboriously to cope with all assigned activities day and night. Time management, therefore, becomes a practical tool for nurse student to reach her goal. It has many good aspects; namely, problem analysis, target determination, planning, implementation, evaluation and revision for improvement .

However, many factors act as barriers to nurse students' attaining and maintaining a high grade point average (GPA) at their training. Faculty members target all these issues in developing strategies to improve students' academic performance and learning achievement. As a result, time management would be a solution to solve these problems.

Investigators would like to determine the effect of skills in time management on GPA amongst faculty nursing students. The research questions are as follows:

1. What is the nurse student's competency on Time management?
2. What is the relationship between GPA and Time management skills among faculty nursing students?

ELIGIBILITY:
Inclusion Criteria:

* volunteered nurse anaesthetist students in 1-year training program

Exclusion Criteria:

* none

Ages: 22 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: nurse anaesthetist students
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
nurse student's competency on Time management | 3 months
  relationship between GPA and Time management skills among nurse students

CONTACTS AND LOCATIONS:
Overall Officials: Suchittra Bumrongsawa, BNS, Principal Investigator — Siriraj Hospital
Locations (1):
- Suchittra Bumrongsawa, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No